CLINICAL TRIAL: NCT05025826
Title: Randomized, Double-blind, Multicenter Placebo-controlled Study Evaluating Neurotoxicity in Patients With Metastatic Gastro Intestinal Cancer Taking Phycocare® or Placebo During Oxaliplatin Based Chemotherapy
Brief Title: Study Evaluating Neurotoxicity in Patients With Metastatic Gastro Intestinal Cancer Taking Phycocare® or Placebo During Oxaliplatin Based Chemotherapy
Acronym: PROPERTY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Algosource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC21_0246
Record Dates: First submitted 2021-07-23; First posted 2021-08-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Gastric Cancer
Keywords: Oxaliplatin based chemotherapy; neurotoxicity
MeSH Terms: conditions — Stomach Neoplasms; Neurotoxicity Syndromes

STUDY DESIGN:
Intervention Model Description: Arm A: Phycocare Arm B: Placebo
Who Masked: Participant, Care Provider
Masking Description: The placebo will match as much as possible all the characteristics of the Phycocare®
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phycocare (Experimental): PHYCOCARE during 12 cycles of 14 days from day -3 before oxaliplatin based chemotherapy until cycle 3 months after the last dose of oxaliplatin (18 cycles, about 9 months) From D-3 to D14 before cycle 1 chemotherapy: patient will take Phycocare From D1 to D14 of cycle 2 chemotherapy and further chemotherapy cycles : patient will take Phycocare On days of chemotherapy the patient does not take Phycocare
  Interventions: Other: Phycocare
- Placebo (Placebo Comparator): Placebo during 12 cycles of 13 days from day -3 before cycle 1 of oxaliplatin based chemotherapy until 3 months after the last dose of oxaliplatin (9 months).
  From D-3 to D13 before cycle 1 chemotherapy: patient will take Placebo From D1 to D13 of cycle 2 chemotherapy and further chemotherapy cycles : patient will take Placebo.
  On days of chemotherapy the patient does not take Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Phycocare — Phycocare every day during 9 months (except days of chemotherapy: no Phycocare)
  Arms: Phycocare
Other: Placebo — Placebo every day during 9 months (except days of chemotherapy = no Placebo)
  Arms: Placebo

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most frequent side effects caused by antineoplastic agents, with a prevalence from 19% to over 85%. Clinically, CIPN is a mostly sensory neuropathy that may be accompanied by motor and autonomic changes of varying intensity and duration.

Due to its high prevalence among cancer patients, CIPN constitutes a major problem for both cancer patients and survivors as well as for their health care providers, especially because, at the moment, there is no single effective method of preventing CIPN; moreover, the possibilities of treating this syndrome are very limited.

The phycocyanin (PC), a biliprotein pigment and an important constituent of the blue-green alga Spirulina platensis, has been reported to possess significant antioxidant and radical-scavenging properties, offering protection against oxidative stress.

Study hypothesis is that phycocyanin may give protection against oxaliplatin-induced neuropathy in the treatment of gastro intestinal cancers including oesogastric, colo-rectal and pancreatic cancers. This trial will be a randomised placebo-controlled study.

DETAILED DESCRIPTION:
The phycocyanin used in this protocol (Phycocare®) will be 5 times more concentrated than the Spirulysat (food supplement commercialized by Algosource).

It will be administrated during Oxaliplatin based chemotherapy and 3 months after oxaliplatin stopped.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with the age > or = to 18 years old.
* Negative pregnancy test for women with child-bearing potential if applicable (without hysterectomy for example)
* Information given to the patient who must have signed informed consent
* Patient with Histologically or cytologically proven gastro intestinal cancer including oesogastric, colo-rectal, pancreatic cancers, locally advanced pancreatic cancers and planned to be treated with oxaliplatin
* Patient with metastatic disease not previously treated
* Patient willing not to take any plant-based therapy during the study (including phytotherapy and gemmotherapy)
* Previous radiotherapy is authorized if discontinued ≥15 days prior to randomization
* Sites of disease evaluated within 42 days prior C1 day 1 of chemotherapy with thoracic-abdominal-pelvic CT scan (or abdominal-pelvic MRI and chest X-ray)
* Patient with ECOG Performance status 0 or 1
* Patients with a Life expectancy ≥12 weeks
* Laboratory results:

Hematologic function:

polynuclear neutrophils ≥ 1.5.109/L platelets ≥100.109/L haemoglobin ≥9 g/dL

Hepatic function:

transaminases ≤2.5 times upper limit of normal (ULN) (≤5 ULN in case of hepatic metastases), alkaline phosphatases ≤2.5 x ULN (≤5 ULN in case of hepatic metastases), total bilirubin ≤1.5 x ULN

Renal function:

creatinemia clearance >50 ml/min (Cockcroft and Gault)

- Patient with Public Health insurance coverage

Exclusion Criteria:

* Patients with phenylketonuria
* Patients with known meningeal or brain metastases
* Patient previously treated for their metastatic cancer
* Patient previously treated with oxaliplatin
* Patient with specific contraindication or known hypersensitivity to spirulina
* Patient with specific contraindication or known hypersensitivity to oxaliplatin.
* Known allergy or hypersensitivity to antibodies or any preservatives if patient is treated with a monoclonal antibody combined to chemotherapy (bevacizumab or cetuximab or panitumumab or nivolumab or Trastuzumab For patients treated with trastuzumab : patient without HER2 overexpression (defined by positive IHC3 or positive IHC2 and confirmed by a positive FISH result)
* Patient with clinically significant coronaries affection or myocardial infarction within 6 months prior to randomization.
* Patient with peripheral neuropathy >1 (CTCAE scale version 5.0).
* Patients with known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Patient with acute intestinal obstruction or sub-obstruction, history of inflammatory intestinal disease or extended resection of the small intestine or presence of a colic prosthesis.
* Patient with unhealed wound, active oesogastric or duodenal ulcer, or bone fracture
* Patient with an history of abdominal fistulas, trachea-esophageal fistulas or any other grade 4, gastro-intestinal perforations or non-gastrointestinal fistulas or intra-abdominal abscesses during the 6 months before randomization.
* For patient treated with bevacizumab: patient with uncontrolled arterial hypertension (systolic pressure >150 mmHg and/or diastolic pressure >100 mmHg) with and without antihypertensive medication. Patients with high hypertension are eligible if antihypertensive medication lowers their arterial pressure to the level specified by the criterion.
* Patient with an history of hypertensive crisis or hypertensive encephalopathy
* Patient with other concomitant malignancy or history of cancer (except in situ carcinoma of the cervix, or non-melanoma skin cancer, treated with curative intent treatment) except if considered in complete remission for at least 2 years before randomization
* Existence of any other pathology, metabolic problem, anomaly during the clinical examination or biological anomaly which may reasonable suspect an underlying pathology which would contra- indicate the use of the study medication or any other risk of complication related to the treatment.
* Any treatment including an experimental drug, or participation in another clinical trial within 28 days before randomization.
* Pregnant women, or women who could possibly be pregnant (or who expect to fall pregnant within 6 months of the end of treatment), or who are breast feeding are not eligible.
* Men and women of child-bearing potential who do not accept to use a highly effective contraceptive (as per currently acceptable institutional standards) or abstinence during the study and for the month after the last administration of the study treatments.
* Persons deprived of liberty or under guardianship.
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Demonstrate a 50% decrease of the grade> or = 2 neurotoxicity at 4 months after oxaliplatin-based chemotherapy start in the PHYCOCARE arm | 4 months after oxaliplatin-based chemotherapy start
  neurotoxicity according to NCI (National Cancer Institute) criteria in both arms

SECONDARY OUTCOMES:
Comparison between the two arms of percentage of patients who stopped oxaliplatin for neurological toxicity | last day of chemotherapy
  Delay of definitive interruption or decrease of oxaliplatin treatment
Comparison between the two arms of percentage of patients with oxaliplatin dose decrease | last day of chemotherapy
  Dose intensity of oxaliplatin
Comparison between the two arms of Neurological toxicities according to the Common Terminology Criteria for adverse Event (CTCAE) v5.0 | end of study visit (an average of 9 months after cycle 1 day1)
  Neurological AE at following hospital visit : baseline, M4 and M9/end of study visit
Comparison between the two arms of Overall Toxicity (including hematological toxicity, gastro-intestinal toxicity, etc…) | end of study visit (an average of 9 months after cycle 1 day1)
  Adverse events grade 1 to 4
Comparison between the two arms of Patient 's Quality of Life according with EORTC-QLQ-C30 | end of study visit (an average of 9 months after cycle 1 day1)
  QLQ C30 - score questions 1 to 28: score frame [30-114] . 30= good quality of life questions 29 and 30 : score frame [2-14] . 2 = bad quality of lifre
Comparison between the two arms of Neurological toxicities | end of study visit (an average of 9 months after cycle 1 day1)
  ElectroNeuroMyography (ENMG) and neurology questionnaire ONLS (overall neuropathy limitations scale)
  ONLS score:
  * sub-score upper limbs : [0-5] . 5= worst neuropathic injury
  * sub score lower limbs [0-7]: 7= worst neuropathic injury
  * total score = upper limbs score + lower limbs score [0-12] ; 0= no injury; 12= maximal incapacity

CONTACTS AND LOCATIONS:
Overall Officials: Yann TOUCHEFEU, Professor, Principal Investigator — NANTES UH
Locations (8):
- France (8):
  - Clermont-Ferrand UH, Clermont-Ferrand, France
  - Centre Hospitalier de Cholet, Cholet
  - Chd La Roche Sur Yon, La Roche-sur-Yon
  - Hôpital le Confluent, Nantes
  - Nantes Uh, Nantes
  - Saint Gregoire Clinique, Rennes
  - Mutaliste Clinic Saint Nazaire, Saint-Nazaire
  - Foch Suresnes Hosptial, Suresnes

REFERENCES:
- [Derived] Le Gouill-Jaijarat C, Pereon Y, Leroy M, Lepine O, Loloum A, Peluchon C, Volteau C, Martineau AS, Korner S, Perrault C, Benmaziane A, Girot P, Petorin C, Perret C, Ligeza-Poisson C, Mayeur D, Flet L, Chiffoleau A, Poinas A, Bennouna J. PROPERTY: study protocol for a randomized, double-blind, multicenter placebo-controlled trial assessing neurotoxicity in patients with metastatic gastrointestinal cancer taking PHYCOCARE(R) during oxaliplatin-based chemotherapy. Trials. 2023 Jan 20;24(1):50. doi: 10.1186/s13063-023-07071-z. PMID 36670495